CLINICAL TRIAL: NCT05284032
Title: A Pilot Trial Using Isatuximab to Overcome Platelet Transfusion Refractoriness in Human Leukocyte Antigen Allo-Immunized Patients
Brief Title: A Pilot Trial Using Isatuximab to Overcome Platelet Transfusion Refractoriness in Human Leukocyte Antigen Allo-Immunized Patients (SuppCare 001)
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Firas El Chaer, MD (Other)
Responsible Party: Sponsor-Investigator, Firas El Chaer, MD, Assistant Professor, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HSR210463
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Platelet Refractoriness; Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Isatuximab (Sarclisa) (Experimental): 4 weekly doses of isatuximab
  Interventions: Drug: isatuximab 10 mg/kg

INTERVENTIONS:
Drug: isatuximab 10 mg/kg — Given by intravenous infusion

SUMMARY:
Some of the treatments for cancer can cause platelets (the part of the blood that helps with clotting) to decrease. If they are too low, then clinicians may recommend a transfusion (getting platelets from another person added to someone else's body). This usually works to increase the person's platelets to a healthy level, but sometimes it doesn't work. This is called platelet refractoriness. This study is trying to find out whether isatuximab (the study drug) may help people with a certain type of platelet refractoriness by removing some cells in order to make platelet transfusions more effective.

DETAILED DESCRIPTION:
Participants in this study will receive 4 weekly infusions of the study drug, isatuximab, by intravenous infusion. The dose of isatuximab infusions may be larger or smaller and take a longer or shorter time to infuse depending on your weight and time required will decrease from the first to second infusion and from the second to third and fourth infusion. Participants will be observed for 2 hours after each infusion. Participants will continue to receive platelet transfusions according to standard clinical care and will be followed for about 120 days after their last dose of isatuximab.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, age ≥ 18 years
4. Diagnosis of immune mediated platelet transfusion refractoriness secondary to class I anti-HLA antibodies according to institutional practice, including calculated percent panel-reactive antibodies (%PRA) > 80%
5. Adequate Organ Function:

   * serum creatinine <= 1.5 x upper limit of normal
   * bilirubin <= 1.5 x upper limit of normal (exceptions for Gilbert's disease)
   * AST and ALT <= 2.5 x upper limit of normal
   * Alkaline phosphatase <= 2.5 x upper limit of normal
6. For females and males of reproductive potential: agreement to use adequate contraception (see section 5.3)
7. Agreement to adhere to Lifestyle Considerations (see Section 5.3) throughout study duration

Exclusion Criteria:

1. Immune-mediated platelet refractoriness other than anti-HLA antibody-mediated
2. Non-immune-mediated platelet refractoriness (e.g. splenomegaly or disseminated intravascular coagulation)
3. Diagnosis of thrombocytopenia induced by other drugs, such as vancomycin, heparin, or amphotericin
4. Diagnosis of thrombotic thrombocytopenic purpura or idiopathic immune thrombocytopenia
5. Active bleeding
6. Greater than Grade 2 active graft versus host disease (GVHD) following allogeneic HSCT
7. Bi-directional ABO mismatched allogeneic stem cell transplantation
8. Prior administration of daratumumab, isatuximab or any other anti-CD38 antibodies
9. Known uncontrolled HIV disease and/or active Hepatitis A, B, or C infection
10. Active systemic infection and severe infections requiring treatment with a parenteral administration of antimicrobials.

    * Controlled systemic infections on antimicrobial therapy that are stable at the time of screening are not an exclusion criterion.
11. Hypersensitivity or history of intolerance to steroids, mannitol, pregelatinized starch, sodium stearyl fumarate, histidine (as base and hydrochloride salt), arginine hydrochloride, poloxamer 188, sucrose or any of the other components of study intervention that are not amenable to premedication with steroids and H2 blockers or would prohibit further treatment with these agents.
12. Received any investigational drug within 14 days or 5 half-lives of the investigational drug prior to initiation of study intervention, whichever is longer. In case of very aggressive disease (i.e acute leukemia) delay could be shortened after agreement between sponsor and investigator, in absence of residual toxicities from previous therapy
13. Pregnancy or lactation
14. Any clinically significant, uncontrolled medical conditions that, in the Investigator's opinion, would expose the patient to excessive risk or may interfere with compliance or interpretation of the study results.
15. Current receipt of, or expectation to require anti-CD20 therapy, proteasome inhibitors, intravenous immune globulin ("IVIG"), and plasma exchange therapy during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Percent panel-reactive antibodies (PRAs)- change over time/with study treatment | Through about 120 days following last study drug infusion
  A weighted percent of class I HLA targets to which the patient has made antibodies

SECONDARY OUTCOMES:
Mean fluorescence intensity (MFI) - change over time/ with study treatment | Through about 120 days following last study drug infusion
  MFI of each class I anti-HLA antibody contributing to the %PRA
Quality of life - changes over time/with study treatment according to the Functional Assessment of Cancer Therapy - Leukemia (FACT-Leu) | Through about 120 days following last study drug infusion
  Each question is scored on a 5-point scale (0 - 4), with a mixture of questions scored with low numbers indicating better quality of life and others indicating worse quality
Adverse events | Through about 30 days following last study drug infusion
  Frequency, severity (by CTCAE v5), and duration of Grade 3 or higher adverse events considered related to the study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Firas El Chaer, MD, Principal Investigator — UVA
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No